CLINICAL TRIAL: NCT04857645
Title: A Phase II Prospective Study "GFM-DACORAL-DLI" ASTX727 and Donor Lymphocyte Infusions After Allogenic Stem Cell Transplantation in Very High Risk MDS or AML Patients
Brief Title: ASTX727 and Donor Lymphocyte Infusions After Allogenic Stem Cell Transplantation in Very High Risk MDS or AML Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-DACORAL-DLI
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: MDS; AML
Keywords: Very high risk MDS; AML; ASTX727; DLI
MeSH Terms: interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASTX727 treatment (Experimental)
  Interventions: Drug: ASTX727; Other: Donor Lymphocyte Infusions

INTERVENTIONS:
Drug: ASTX727 — Eligible patient started ASTX727 between 40 and 130 days after allogenic stem cell transplantation
Other: Donor Lymphocyte Infusions — In absence of previous grade 2-4 or chronic graft-versus-host disease (GVHD), DLI will be administered at increasing doses the first day of ASTX727 cycles
  Other Names: DLI

SUMMARY:
Study of early administration of ASTX727 associated with late Donor Lymphocyte Infusions after allogenic stem cell transplantation in very high risk MDS or AML patients

DETAILED DESCRIPTION:
Prospective study of early administration of ASTX727 associated with late Donor Lymphocyte Infusions after allogenic stem cell transplantation in very high risk MDS or AML patients

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 70 years
* MDS or AML with unfavorable genetics defined as follow:
* 4 or more cytogenetic abnormalities or
* 3 cytogenetic abnormalities and TP53 or other unfavorable mutations (ASXL1, RUNX1) or
* 3 cytogenetic abnormalities and monosomal karyotype or
* mutations involving EVI1
* AML patients should have received chemotherapy
* Marrow blast < 20% for MDS and < 10% for AML post chemotherapy
* For MDS : Revised IPSS poor or very poor ; For AML : ELN adverse risk
* Non-proliferative disease
* A donor is available (HLA matched or mismatched)
* Adequate contraception in women < 50 years and for men. Subjects must agree to use, and to be able to comply with, effective contraception without interruption, at least the first six months after transplant, throughout the entire duration of study drug therapy and for at least 6 months for women and 3 months for men after the last dose of study drug therapy.

Exclusion Criteria:

* ECOG 3 or more
* Cancer less than 2 years before inclusion or cancer not in remission the last 2 years before inclusion (except in situ cancer or baso cellular cancer)
* Cardiac failure with Ejection Fraction < 50%
* Creatininemia level > 150 µmol/L
* Liver enzyme > 3 N
* Conjugated bilirubinemia > 25 µmol/L
* MDS occurring in patients with Fanconi anemia or congenital dyskeratosis
* Proliferative disease in patients not in remission: White Blood Cell (WBC) > 15 G/L or use of continuous cytotoxic to maintain WBC < 15 G/L
* AML with marrow or peripheral blast count higher than 10% after chemotherapy
* Known allergy or hypersensitivity to the investigational agent or decitabine or its metabolites or formulation excipients
* No contraception
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Disease free Survival (DFS) at one year post transplant | 1 year post transplant
  Measure of time during which no sign of progression is found

SECONDARY OUTCOMES:
Overall Survival (OS) at one year post transplant | 1 year post transplant
  Measure of time from randomization to death from any cause
Overall Survival (OS) at two years post transplant | 2 years post transplant
  Measure of time from randomization to death from any cause
Risk factors for DFS, OS and non-relapse mortality at 1 and 2 years | 1 and 2 years
  Statistical study of cumulative incidence curves

CONTACTS AND LOCATIONS:
Overall Officials: Marie ROBIN, MD, Principal Investigator — Hôpital Saint Louis - Service hématologie-greffe; Pierre FENAUX, MD, Principal Investigator — Hôpital Saint Louis - Service hématologie séniors
Locations (12):
- France (12):
  - CHU d'Amiens Picardie - Site sud - Service hématologie clinique et thérapie cellulaire, Amiens
  - CHU d'Angers - Service des maladies du sang, Angers
  - CHU Estaing - Service hématologie clinique et thérapie cellulaire, Clermont-Ferrand
  - CHU de Grenoble - Clinique Universitaire d'hématologie, Grenoble
  - Hôpital Saint Eloi - Service hématologie clinique, Montpellier
  - CHU Hôtel Dieu - Service hématologie clinique, Nantes
  - Hôpital Saint Louis - Service hématologie-greffe, Paris
  - CHU de Haut-Lévèque de Bordeaux - Service des maladies du sang, Pessac
  - CH Lyon Sud - Servide Hématologie, Pierre-Bénite
  - Centre Henri Becquerel - Département d'hématologie, Rouen
  - IUCT Oncopole - Département d'hématologie - Service de greffe de cellules souches hématopoïétiques, Toulouse
  - CHU Brabois - Service hématologie clinique, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robin M, D'Aveni M, Stamatoullas A, Raffoux E, Chevallier P, Garnier A, Mediavilla C, Carre M, Himberlin C, Sebert M, Ravinet A, Desseaux K, Labussiere H, Alani M, Rubio MT, Huynh A, Ades L, de Latour RP, Paul F, Chermat F, Petit R, Mokeddem C, Charbonnier A, Thepot S, Chevret S, Fenaux P; Societe Francophone de Greffe de Moelle et de Therapie Cellulaire (SFGM-TC) and the Groupe Francophone des Myelodysplasies (GFM). Oral decitabine and cedazuridine maintenance after haematopoietic stem-cell transplantation in very high-risk acute myeloid leukaemia or myelodysplastic syndrome (GFM-DACORAL-DLI): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2025 Sep;12(9):e705-e716. doi: 10.1016/S2352-3026(25)00172-3. Epub 2025 Aug 7. PMID 40784355